CLINICAL TRIAL: NCT04922281
Title: Insertable Cardiac Monitor-Guided Early Intervention to Reduce Atrial Fibrillation Burden Following Catheter Ablation (ICM REDUCE-AF)
Brief Title: Insertable Cardiac Monitor-Guided Early Intervention to Reduce Atrial Fibrillation Burden Following Catheter Ablation
Acronym: ICMREDUCE-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ilan Goldenberg, Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00005723; R61HL153001 (NIH)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac; Pathologic Processes
Keywords: ICM, Confirm Rx™ , AF Ablation, Atrial Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac; Pathologic Processes | interventions — Complementary Therapies

STUDY DESIGN:
Intervention Model Description: The study population will include 120 subjects with history of paroxysmal or persistent AF who have been referred for a CA procedure based on conventional clinical indications and who will be randomized 1:1 to conventional (control arm) or ICM/CIED/non-invasive LT-ECG monitor-guided management (early intervention arm).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Physicians and subjects will be blinded to SCAF detected by the ICM/CIED/non-invasive LT-ECG monitor, but will be provided by the DCC upon request with full ICM/CIED/non-invasive LT-ECG monitor information on any clinical episodes. Cause-specific hospitalization and ED will be adjudicated by an independent and blinded Events Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ICM/CIED/non-invasive LT-ECG patch arrhythmia detection guided Management (Active Comparator): Implantable device (ICM/CIED) that provides accurate daily transmission of cardiac electrical data for arrhythmia detection. Patients without an existing CIED who prefer to use noninvasive LT-ECG monitoring will be offered to use the Carnation Ambulatory Monitor ("CAM™"; Bardy Diagnostics). The CAM™ is patch approved for LT-ECG monitoring applied to the skin over the chest for a time-period of 7-days every 2 months for cardiac electrical data for arrhythmia detection.
  Interventions: Device: Insertable Cardiac Monitor or external non-invasive LT-ECG patch
- Conventional Management (Placebo Comparator): Treating physicians/nurses will be blinded to the AF episodes data from the monitor, but will be provided information on asystole, or ventricular arrhythmia events (for safety).
  Interventions: Device: Insertable Cardiac Monitor or external non-invasive LT-ECG patch

INTERVENTIONS:
Device: Insertable Cardiac Monitor or external non-invasive LT-ECG patch — Implantable device that provides accurate daily transmission. Patients without an existing CIED who prefer to use noninvasive LT-ECG monitoring will be offered to use the Carnation Ambulatory Monitor ("CAM™"; Bardy Diagnostics) the CAM™ patch approved for LT-ECG monitoring applied to the skin over the chest for a time-period of 7-days every 2 months for cardiac electrical data for arrhythmia detection.
  Other Names: Confirm Rx™; Carnation Ambulatory Monitor ("CAM™"; Bardy Diagnostics).The CAM™ patch.

SUMMARY:
To prospectively investigate the efficacy of an insertable cardiac monitor-guided atrial fibrillation (AF) management in reducing subsequent AF burden in patients with persistent or paroxysmal AF undergoing atrial catheter ablation (CA).

DETAILED DESCRIPTION:
In this study, 120 subjects from the University of Rochester enrolling site will be randomized (1:1) to conventional AF management vs. Abbott ICM- guided AF management following ablation for persistent AF. Subjects will be followed for 15 months including a 3 month blanking period following AF ablation. The study subject population will include subjects with paroxysmal atrial fibrillation (per 2019 HRS guidelines definition: an episode of AF that terminates spontaneously or with intervention in less than seven days) or persistent atrial fibrillation (sustained AF episode lasting more than 7 days, but less than 1 year), according to current guideline indications for persistent AF ablation and Abbott ICM implantation. The Abbott ICM incorporates a mobile app (myMerlin) that allows early detection of AF recurrence through patient-triggered remote transmissions and correlation with symptoms based on subclinical AF (SCAF) and patient-triggered remote transmissions. Future FDA-approved Abbott ICM devices using the same functionality may also be utilized in this study. This is a Phase 4 study, and we are comparing two management strategies that are currently employed in clinical practice.

ELIGIBILITY:
Inclusion criteria

* History of paroxysmal atrial fibrillation (per 2019 HRS guidelines definition: an episode of AF that terminates spontaneously or with intervention in less than seven days), according to current guideline indications for paroxysmal AF CA (Class I/II); or patients with history of persistent atrial fibrillation (per 2019 HRS guidelines definition: sustained AF episode lasting more than 7 days, but less than 3 years), according to current guideline indications for persistent AF CA (Class I/IIIa) any time in the past.
* 18 years of age or older at time of consent
* CA to be performed for AF as standard of care within 2 calendar months after consent and prior to randomization date
* One of the following:

  * Abbott ICM device indicated for monitoring symptoms after CA as standard of care and inserted within 2 calendar months after consent and prior to randomization date
  * Patients with an existing CIED (ICD/CRTD/PPM/ICM) are allowed if there is an atrial lead to track AF.
  * Patient without an existing CIED preferring to use a noninvasive LT-ECG monitor.

Exclusion criteria

* Inability or unwilling to undergo CA (e.g., presence of intra-cardiac thrombus, contraindication to anticoagulation or other contraindication to CA)
* Inability to tolerate any AAD therapy
* Permanent atrial fibrillation lasting more than 3 years prior to date of consent
* NYHA class IV congestive heart failure
* Life expectancy <1 year after consent date for any medical condition
* Pregnancy or nursing
* Unwillingness to comply with all post-procedural follow-up requirements and to sign informed consent
* Participation in other interventional research studies (observational registries are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean amount of time spent in AF | 3-15 months (12 months)
  The primary endpoint of the trial is total AF burden between 3 and 15 months after the index CA procedure (i.e. over 1-year post-blanking), as detected by an ICM which will be inserted prior to or at the time of the CA procedure, existing CIED, or non-invasive LT-ECG monitor in all study subjects. AF recurrence is defined as any episode of AF lasting >30 seconds. AF burden will be defined as the mean amount of time spent in AF over the pre-specified period of time (excluding short AF episodes of ≤30 seconds).

SECONDARY OUTCOMES:
Mean Healthcare utilization | 15 months
  Total number of hospitalizations for any cause, ED visits, and unplanned office visits recorded at each study follow-up visit
Mean change in Functional capacity as measured by Cardiopulmonary Exercise Test (CPET) | Baseline to 15 months
  Function capacity will be reported as peak VO2, which will be determined from CPET.
Mean change in Functional capacity as measured by ICM | Baseline to 15 months
  The average daily count of steps derived from the inserted cardiac monitor
Mean change in Quality of life using the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) questionnaire | Baseline to 15 months
  The AFEQT questionnaire will be used to collect quality of life data. The questionnaire has 20 questions on a 7-point Likert scale that assess symptoms, daily activities and treatment concerns. Scores range from 20-140 with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Writing Group Members; January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS focused update of the 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Heart Rhythm. 2019 Aug;16(8):e66-e93. doi: 10.1016/j.hrthm.2019.01.024. Epub 2019 Jan 28. No abstract available. PMID 30703530
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Kim MH, Johnston SS, Chu BC, Dalal MR, Schulman KL. Estimation of total incremental health care costs in patients with atrial fibrillation in the United States. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):313-20. doi: 10.1161/CIRCOUTCOMES.110.958165. Epub 2011 May 3. PMID 21540439
- [Background] Terasawa T, Balk EM, Chung M, Garlitski AC, Alsheikh-Ali AA, Lau J, Ip S. Systematic review: comparative effectiveness of radiofrequency catheter ablation for atrial fibrillation. Ann Intern Med. 2009 Aug 4;151(3):191-202. doi: 10.7326/0003-4819-151-3-200908040-00131. Epub 2009 Jul 6. PMID 19581635
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Arbelo E, Brugada J, Hindricks G, Maggioni AP, Tavazzi L, Vardas P, Laroche C, Anselme F, Inama G, Jais P, Kalarus Z, Kautzner J, Lewalter T, Mairesse GH, Perez-Villacastin J, Riahi S, Taborsky M, Theodorakis G, Trines SA; Atrial Fibrillation Ablation Pilot Study Investigators. The atrial fibrillation ablation pilot study: a European Survey on Methodology and results of catheter ablation for atrial fibrillation conducted by the European Heart Rhythm Association. Eur Heart J. 2014 Jun 7;35(22):1466-78. doi: 10.1093/eurheartj/ehu001. Epub 2014 Jan 31. PMID 24487524
- [Background] Kuck KH, Hoffmann BA, Ernst S, Wegscheider K, Treszl A, Metzner A, Eckardt L, Lewalter T, Breithardt G, Willems S; Gap-AF-AFNET 1 Investigators*. Impact of Complete Versus Incomplete Circumferential Lines Around the Pulmonary Veins During Catheter Ablation of Paroxysmal Atrial Fibrillation: Results From the Gap-Atrial Fibrillation-German Atrial Fibrillation Competence Network 1 Trial. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003337. doi: 10.1161/CIRCEP.115.003337. PMID 26763226
- [Background] Hosseini SM, Rozen G, Saleh A, Vaid J, Biton Y, Moazzami K, Heist EK, Mansour MC, Kaadan MI, Vangel M, Ruskin JN. Catheter Ablation for Cardiac Arrhythmias: Utilization and In-Hospital Complications, 2000 to 2013. JACC Clin Electrophysiol. 2017 Nov;3(11):1240-1248. doi: 10.1016/j.jacep.2017.05.005. Epub 2017 Aug 2. PMID 29759619
- [Background] Calkins H, Reynolds MR, Spector P, Sondhi M, Xu Y, Martin A, Williams CJ, Sledge I. Treatment of atrial fibrillation with antiarrhythmic drugs or radiofrequency ablation: two systematic literature reviews and meta-analyses. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):349-61. doi: 10.1161/CIRCEP.108.824789. Epub 2009 Jun 2. PMID 19808490
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Darkner S, Chen X, Hansen J, Pehrson S, Johannessen A, Nielsen JB, Svendsen JH. Recurrence of arrhythmia following short-term oral AMIOdarone after CATheter ablation for atrial fibrillation: a double-blind, randomized, placebo-controlled study (AMIO-CAT trial). Eur Heart J. 2014 Dec 14;35(47):3356-64. doi: 10.1093/eurheartj/ehu354. Epub 2014 Sep 2. PMID 25182250
- [Background] Verma A, Kilicaslan F, Pisano E, Marrouche NF, Fanelli R, Brachmann J, Geunther J, Potenza D, Martin DO, Cummings J, Burkhardt JD, Saliba W, Schweikert RA, Natale A. Response of atrial fibrillation to pulmonary vein antrum isolation is directly related to resumption and delay of pulmonary vein conduction. Circulation. 2005 Aug 2;112(5):627-35. doi: 10.1161/CIRCULATIONAHA.104.533190. PMID 16061753
- [Background] Callans DJ, Gerstenfeld EP, Dixit S, Zado E, Vanderhoff M, Ren JF, Marchlinski FE. Efficacy of repeat pulmonary vein isolation procedures in patients with recurrent atrial fibrillation. J Cardiovasc Electrophysiol. 2004 Sep;15(9):1050-5. doi: 10.1046/j.1540-8167.2004.04052.x. PMID 15363079
- [Background] Nanthakumar K, Plumb VJ, Epstein AE, Veenhuyzen GD, Link D, Kay GN. Resumption of electrical conduction in previously isolated pulmonary veins: rationale for a different strategy? Circulation. 2004 Mar 16;109(10):1226-9. doi: 10.1161/01.CIR.0000121423.78120.49. Epub 2004 Mar 1. PMID 14993124
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] Lellouche N, Jais P, Nault I, Wright M, Bevilacqua M, Knecht S, Matsuo S, Lim KT, Sacher F, Deplagne A, Bordachar P, Hocini M, Haissaguerre M. Early recurrences after atrial fibrillation ablation: prognostic value and effect of early reablation. J Cardiovasc Electrophysiol. 2008 Jun;19(6):599-605. doi: 10.1111/j.1540-8167.2008.01188.x. Epub 2008 May 5. PMID 18462321
- [Background] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Turov A, Shirokova N, Karaskov A. Use of an implantable monitor to detect arrhythmia recurrences and select patients for early repeat catheter ablation for atrial fibrillation: a pilot study. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):823-31. doi: 10.1161/CIRCEP.111.964809. Epub 2011 Sep 19. PMID 21930653
- [Background] Alipour P, Azizi Z, Pirbaglou M, Ritvo P, Pantano A, Verma A, Khaykin Y. Defining Blanking Period Post-Pulmonary Vein Antrum Isolation. JACC Clin Electrophysiol. 2017 Jun;3(6):568-576. doi: 10.1016/j.jacep.2017.01.006. Epub 2017 Mar 29. PMID 29759429
- [Background] Pokushalov E, Romanov A, De Melis M, Artyomenko S, Baranova V, Losik D, Bairamova S, Karaskov A, Mittal S, Steinberg JS. Progression of atrial fibrillation after a failed initial ablation procedure in patients with paroxysmal atrial fibrillation: a randomized comparison of drug therapy versus reablation. Circ Arrhythm Electrophysiol. 2013 Aug;6(4):754-60. doi: 10.1161/CIRCEP.113.000495. Epub 2013 Jun 7. PMID 23748210
- [Background] Eitel C, Husser D, Hindricks G, Fruhauf M, Hilbert S, Arya A, Gaspar T, Wetzel U, Bollmann A, Piorkowski C. Performance of an implantable automatic atrial fibrillation detection device: impact of software adjustments and relevance of manual episode analysis. Europace. 2011 Apr;13(4):480-5. doi: 10.1093/europace/euq511. Epub 2011 Feb 16. PMID 21325346
- [Background] Hindricks G, Piorkowski C, Tanner H, Kobza R, Gerds-Li JH, Carbucicchio C, Kottkamp H. Perception of atrial fibrillation before and after radiofrequency catheter ablation: relevance of asymptomatic arrhythmia recurrence. Circulation. 2005 Jul 19;112(3):307-13. doi: 10.1161/CIRCULATIONAHA.104.518837. Epub 2005 Jul 11. PMID 16009793
- [Background] Ziegler PD, Koehler JL, Mehra R. Comparison of continuous versus intermittent monitoring of atrial arrhythmias. Heart Rhythm. 2006 Dec;3(12):1445-52. doi: 10.1016/j.hrthm.2006.07.030. Epub 2006 Aug 3. PMID 17161787
- [Background] Lewalter T, Boriani G. Relevance of Monitoring Atrial Fibrillation in Clinical Practice. Arrhythm Electrophysiol Rev. 2012 Sep;1(1):54-58. doi: 10.15420/aer.2012.1.54. PMID 26835031
- [Background] Zuern CS, Kilias A, Berlitz P, Seizer P, Gramlich M, Muller K, Duckheim M, Gawaz M, Schreieck J. Anticoagulation after catheter ablation of atrial fibrillation guided by implantable cardiac monitors. Pacing Clin Electrophysiol. 2015 Jun;38(6):688-93. doi: 10.1111/pace.12625. Epub 2015 Apr 13. PMID 25753968
- [Background] Verma A, Champagne J, Sapp J, Essebag V, Novak P, Skanes A, Morillo CA, Khaykin Y, Birnie D. Discerning the incidence of symptomatic and asymptomatic episodes of atrial fibrillation before and after catheter ablation (DISCERN AF): a prospective, multicenter study. JAMA Intern Med. 2013 Jan 28;173(2):149-56. doi: 10.1001/jamainternmed.2013.1561. PMID 23266597
- [Background] Pedrote A, Arana-Rueda E, Garcia-Riesco L, Sanchez-Brotons J, Duran-Guerrero M, Gomez-Pulido F, Arce-Leon A, Frutos-Lopez M. Paroxysmal atrial fibrillation burden before and after pulmonary veins isolation: an observational study through a subcutaneous leadless cardiac monitor. J Cardiovasc Electrophysiol. 2013 Oct;24(10):1075-82. doi: 10.1111/jce.12190. Epub 2013 Jun 21. PMID 23790041
- [Background] Tondo C, Tritto M, Landolina M, DE Girolamo P, Bencardino G, Moltrasio M, Dello Russo A, Della Bella P, Bertaglia E, Proclemer A, DE Sanctis V, Mantica M. Rhythm-symptom correlation in patients on continuous monitoring after catheter ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2014 Feb;25(2):154-60. doi: 10.1111/jce.12292. Epub 2013 Oct 21. PMID 24102697
- [Background] Wechselberger S, Kronborg M, Huo Y, Piorkowski J, Neudeck S, Passler E, El-Armouche A, Richter U, Mayer J, Ulbrich S, Pu L, Kirstein B, Gaspar T, Piorkowski C. Continuous monitoring after atrial fibrillation ablation: the LINQ AF study. Europace. 2018 Nov 1;20(FI_3):f312-f320. doi: 10.1093/europace/euy038. PMID 29688326
- [Background] Hohnloser SH, Capucci A, Fain E, Gold MR, van Gelder IC, Healey J, Israel CW, Lau CP, Morillo C, Connolly SJ; ASSERT Investigators and Committees. ASymptomatic atrial fibrillation and Stroke Evaluation in pacemaker patients and the atrial fibrillation Reduction atrial pacing Trial (ASSERT). Am Heart J. 2006 Sep;152(3):442-7. doi: 10.1016/j.ahj.2006.02.016. PMID 16923410
- [Background] Chen LY, Chung MK, Allen LA, Ezekowitz M, Furie KL, McCabe P, Noseworthy PA, Perez MV, Turakhia MP; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Atrial Fibrillation Burden: Moving Beyond Atrial Fibrillation as a Binary Entity: A Scientific Statement From the American Heart Association. Circulation. 2018 May 15;137(20):e623-e644. doi: 10.1161/CIR.0000000000000568. Epub 2018 Apr 16. PMID 29661944
- [Background] Gonzalez M, Keating RJ, Markowitz SM, Liu CF, Thomas G, Ip JE, Lerman BB, Cheung JW. Newly detected atrial high rate episodes predict long-term mortality outcomes in patients with permanent pacemakers. Heart Rhythm. 2014 Dec;11(12):2214-21. doi: 10.1016/j.hrthm.2014.08.019. Epub 2014 Aug 15. PMID 25131667
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- [Background] Pontoppidan J, Nielsen JC, Poulsen SH, Hansen PS. Symptomatic and asymptomatic atrial fibrillation after pulmonary vein ablation and the impact on quality of life. Pacing Clin Electrophysiol. 2009 Jun;32(6):717-26. doi: 10.1111/j.1540-8159.2009.02357.x. PMID 19545333
- [Background] Skalski J, Allison TG, Miller TD. The safety of cardiopulmonary exercise testing in a population with high-risk cardiovascular diseases. Circulation. 2012 Nov 20;126(21):2465-72. doi: 10.1161/CIRCULATIONAHA.112.110460. Epub 2012 Oct 22. PMID 23091065
- [Background] Kim YG, Shim J, Choi JI, Kim YH. Radiofrequency Catheter Ablation Improves the Quality of Life Measured with a Short Form-36 Questionnaire in Atrial Fibrillation Patients: A Systematic Review and Meta-Analysis. PLoS One. 2016 Sep 28;11(9):e0163755. doi: 10.1371/journal.pone.0163755. eCollection 2016. PMID 27681507
- [Background] Kotecha D, Ahmed A, Calvert M, Lencioni M, Terwee CB, Lane DA. Patient-Reported Outcomes for Quality of Life Assessment in Atrial Fibrillation: A Systematic Review of Measurement Properties. PLoS One. 2016 Nov 1;11(11):e0165790. doi: 10.1371/journal.pone.0165790. eCollection 2016. PMID 27802324
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] Ladapo JA, David G, Gunnarsson CL, Hao SC, White SA, March JL, Reynolds MR. Healthcare utilization and expenditures in patients with atrial fibrillation treated with catheter ablation. J Cardiovasc Electrophysiol. 2012 Jan;23(1):1-8. doi: 10.1111/j.1540-8167.2011.02130.x. Epub 2011 Jul 21. PMID 21777324
- [Background] Hunter RJ, Berriman TJ, Diab I, Kamdar R, Richmond L, Baker V, Goromonzi F, Sawhney V, Duncan E, Page SP, Ullah W, Unsworth B, Mayet J, Dhinoja M, Earley MJ, Sporton S, Schilling RJ. A randomized controlled trial of catheter ablation versus medical treatment of atrial fibrillation in heart failure (the CAMTAF trial). Circ Arrhythm Electrophysiol. 2014 Feb;7(1):31-8. doi: 10.1161/CIRCEP.113.000806. Epub 2014 Jan 1. PMID 24382410
- [Background] Fleiss JL. Analysis of data from multiclinic trials. Control Clin Trials. 1986 Dec;7(4):267-75. doi: 10.1016/0197-2456(86)90034-6. PMID 3802849
- [Background] Hilgers RD, Manolov M, Heussen N, Rosenberger WF. Design and analysis of stratified clinical trials in the presence of bias. Stat Methods Med Res. 2020 Jun;29(6):1715-1727. doi: 10.1177/0962280219846146. Epub 2019 May 10. PMID 31074333
- [Background] Xi W, Pennell ML, Andridge RR, Paskett ED. Comparison of intent-to-treat analysis strategies for pre-post studies with loss to follow-up. Contemp Clin Trials Commun. 2018 May 9;11:20-29. doi: 10.1016/j.conctc.2018.05.008. eCollection 2018 Sep. PMID 30023456
- [Background] Huque MH, Carlin JB, Simpson JA, Lee KJ. A comparison of multiple imputation methods for missing data in longitudinal studies. BMC Med Res Methodol. 2018 Dec 12;18(1):168. doi: 10.1186/s12874-018-0615-6. PMID 30541455
- [Background] Beinart SC, Natale A, Verma A, Amin A, Kasner S, Diener HC, Pouliot E, Franco N, Mittal S. Real-World Use of Prophylactic Antibiotics in Insertable Cardiac Monitor Procedures. Pacing Clin Electrophysiol. 2016 Aug;39(8):837-42. doi: 10.1111/pace.12886. Epub 2016 Jun 7. PMID 27198480
- [Background] Schmidt M, Dorwarth U, Andresen D, Brachmann J, Kuck KH, Kuniss M, Lewalter T, Spitzer S, Willems S, Senges J, Junger C, Hoffmann E. Cryoballoon versus RF ablation in paroxysmal atrial fibrillation: results from the German Ablation Registry. J Cardiovasc Electrophysiol. 2014 Jan;25(1):1-7. doi: 10.1111/jce.12267. Epub 2013 Oct 17. PMID 24134539
- [Background] Hindricks G, Pokushalov E, Urban L, Taborsky M, Kuck KH, Lebedev D, Rieger G, Purerfellner H; XPECT Trial Investigators. Performance of a new leadless implantable cardiac monitor in detecting and quantifying atrial fibrillation: Results of the XPECT trial. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):141-7. doi: 10.1161/CIRCEP.109.877852. Epub 2010 Feb 16. PMID 20160169
- [Background] Gerstenfeld EP, Callans DJ, Dixit S, Zado E, Marchlinski FE. Incidence and location of focal atrial fibrillation triggers in patients undergoing repeat pulmonary vein isolation: implications for ablation strategies. J Cardiovasc Electrophysiol. 2003 Jul;14(7):685-90. doi: 10.1046/j.1540-8167.2003.03013.x. PMID 12930245